CLINICAL TRIAL: NCT01936922
Title: Testing Whether Brief Use of a Wearable Virtual Reality Device Improves Gait, Balance, and Confidence After Falls
Brief Title: Testing Whether Brief Use of a Virtual Reality Device Improves Gait
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, Nimali Jayasinghe, Assistant Professor of Psychology, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1303013747
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Falls, Accidental
Keywords: Fall accidents; Gait; Balance; Fear of falling; Virtual reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Virtual reality device (GaitAid®) (Experimental): This will be a within-subjects design. Each subject will first walk in a controlled laboratory setting as she or he would in daily life. After this, each participant will walk while using the virtual reality device (GaitAid®) for a brief period of time. The session will end with walking as usual.
  Interventions: Device: GaitAid®

INTERVENTIONS:
Device: GaitAid® — Provides visual and auditory cues for walking.

SUMMARY:
A virtual reality device has already been successfully used for improving gait in adults who have neurological conditions. We will evaluate if it is feasible to study the brief use of this device in older adults who have had falls.

DETAILED DESCRIPTION:
Older adults are at risk for recurrent falls.

This study will involve a single study session (lasting two hours) in the controlled setting of a research laboratory. This study will evaluate whether older adults who have had unintentional falls are willing to enroll in this kind of study, use the device briefly, and undergo research assessments. The study will also test whether using the virtual reality device leads to detectable changes in gait, balance, and mobility confidence. This study will lay the groundwork for more comprehensive studies in the future that will assess the clinical impact of using the device.

Twenty-four subjects will be recruited. They will include equal numbers of older adults who: (1) have fallen without a significant injury (e.g. only minor contusion, lacerations) or (2) have fallen with a significant injury (e.g. dislocation, strain/sprain, or fracture) which has healed prior to enrollment.

Each subject will complete baseline measures of gait, balance, and confidence. Then she or he will be introduced to the virtual reality device and will use it for a brief period. Gait and balance will be tested again, first with the virtual reality device and then, finally, without the virtual reality device.

The device (GaitAid®), developed by co-investigator Yoram Baram, Ph.D., has already been used for the rehabilitation of neurological patients (e.g. Parkinson's Disease). The device is a training tool and NOT a continuous walking aid.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60+.
2. English-speaking.
3. One or more unintentional falls in past year.
4. Able to ambulate for at least 10 minutes without continuous assistance, i.e., without human physical assistance and without an assistive device such as a walker, or a cane.
5. A moderate or high level of concern about falling (determined by phone screening by PI).
6. Community dwelling.

   Exclusion Criteria:
7. Diagnosed with any neurological disease, i.e., sensory ataxia, cerebellar ataxia, or spasticity of the lower limbs.
8. Diagnosed with Parkinson's Disease.
9. Diagnosed with Multiple Sclerosis.
10. Diagnosed with Cerebral Palsy.
11. Marked cognitive impairment.
12. Uses large eyeglasses to walk.
13. Vision conditions that reduce ability to use the device.
14. Severe hearing loss.
15. Unstable medical condition or terminal illness.
16. Inability to otherwise comply with the study procedures (determined by PI/study clinician).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Step length | Two hours
  Step length will be measured by GaitMat II® at three time points within the single study session: before using the virtual reality device, while using the virtual reality device, and after using the virtual reality device.

SECONDARY OUTCOMES:
Postural Sway | Two hours
  Postural sway will be measured by a plantar pressure measuring device (Novel [Munich, Germany] emed-X) at three time-points during the two-hour study session: before using the virtual reality device, while using the virtual reality device, and again after using the virtual reality device.
Fear of Falling | Two hours
  Fear of falling will be measured using a visual analog scale at three time-points during the two-hour study session: before using the virtual reality device, while using the virtual reality device, and again after using the virtual reality device.
Single support time | Two hours
  Another aspect of gait, single support time, will also be measured by GaitMat II® at three time points within the single study session: before using the virtual reality device, while using the virtual reality device, and after using the virtual reality device.
Walking velocity | Two hours
  Another aspect of gait, walking velocity, will be measured by GaitMat II® at three time points within the single study session: before using the virtual reality device, while using the virtual reality device, and after using the virtual reality device.

CONTACTS AND LOCATIONS:
Overall Officials: Nimali Jayasinghe, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States